CLINICAL TRIAL: NCT05256173
Title: Clinical Study on the Effect of Improving Sleep Quality on Cognitive Function in Patients With Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20212171-F-1
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Epilepsy，Cognition
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Melatonin Tablets (Experimental)
  Interventions: Other: Melatonin Tablets
- Lactasin Tablets (Placebo Comparator)
  Interventions: Other: Lactasin Tablets
- transcutaneous vagus nerve stimulation (Experimental)
  Interventions: Device: transcutaneous vagus nerve stimulation
- sham transcutaneous vagus nerve stimulation (Sham Comparator)
  Interventions: Device: sham transcutaneous vagus nerve stimulation

INTERVENTIONS:
Other: Melatonin Tablets — Melatonin Tablets was given 3 tablets (6.21mg) daily at the beginning of bedtime at night for a total of 4 weeks.
  Arms: Melatonin Tablets
Other: Lactasin Tablets — The placebo group was given at the beginning of bedtime at night for a total of 4 weeks.
  Arms: Lactasin Tablets
Device: transcutaneous vagus nerve stimulation — transcutaneous vagus nerve stimulation treatment, frequency 10Hz, stimulation site is the anterior wall of the left external auditory canal (tragus), used twice a day, each treatment for 30 minutes, a total of 4 weeks.
  Arms: transcutaneous vagus nerve stimulation
Device: sham transcutaneous vagus nerve stimulation — In the sham stimulation group, the stimulation site was the left earlobe with a frequency of 10Hz, which was used twice a day for 30 minutes for a total of 4 weeks.
  Arms: sham transcutaneous vagus nerve stimulation

SUMMARY:
Epilepsy is one of the common chronic diseases of the central nervous system. 30% to 40% of patients with epilepsy have varying degrees of cognitive impairment, which affects their quality of life. At present, the treatment of cognitive impairment in patients with epilepsy is relatively scarce, and the therapeutic effect is still not ideal. Recent studies have shown that sleep disorder is also an important factor causing cognitive dysfunction, and improving sleep quality has a prospect to become a new way to treat cognitive impairment in patients with epilepsy. The purpose of this study is to observe the relationship between sleep and cognitive function in patients with epilepsy, and to improve the sleep quality of patients with epilepsy, so as to provide new ideas for improving cognitive impairment in patients with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* 1. In accordance with the diagnostic criteria of epilepsy; 2. History of epilepsy ≥ 1 year; 3. Epilepsy with cognitive impairment; 4. Age 7-65 years old; 5. There was no change in the type and dose of antiepileptic drugs during the experiment; 6. Patients and their families were aware of this study and signed an informed consent form.

Exclusion Criteria:

* 1. Status epilepticus; 2. Complicated with severe infection, cerebrovascular diseases, malignant tumors, other nervous system diseases, and systemic diseases that can involve the nervous system (such as immune diseases, etc.), serious dysfunction of heart, liver, kidney and other organs; 3. Non-epileptic seizures such as syncope and hysteria; 4. Women during lactation or pregnancy; 5. Combined use of sleeping and sedative drugs; 6. There are contraindications of melatonin and percutaneous vagal nerve stimulation (tVNS).

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | Week 4
  The difference between the end of treatment score and the baseline

SECONDARY OUTCOMES:
Rey complex figure test | Week 4
  The difference between the end of treatment score and the baseline
Rey auditory verbal learning test | Week 4
  The difference between the end of treatment score and the baseline
Boston naming test | Week 4
  The difference between the end of treatment score and the baseline
Quality of life questionnaire in epilepsy inventory | Week 4
  The difference between the end of treatment score and the baseline
Wechsler Memory Scale | Week 4
  The difference between the end of treatment score and the baseline
Pittsburgh sleep quality index | Week 4
  The difference between the end of treatment score and the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital,the Air Force Medical University, Xi'an, Shaanxi, China